CLINICAL TRIAL: NCT04851717
Title: A Phase 2/3, Prospective, Open-label Trial Evaluating the Efficacy, Safety, and Pharmacokinetics of Remimazolam for Intravenous Sedation in Paediatric Patients Undergoing Diagnostic and/or Therapeutic Procedures
Brief Title: Investigation of Remimazolam in Children Undergoing Sedation for Medical Procedures
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Acacia Pharma Ltd (Industry)
Collaborators: Paion UK Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DA10030; CNS7056-026 (Other: PAION)
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — remimazolam

STUDY DESIGN:
Intervention Model Description: A Phase 2/3 prospective, open-label trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All Patients (Experimental): All paediatric patients undergoing diagnostic and/or therapeutic procedures
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — Remimazolam for intravenous sedation

SUMMARY:
To assess the efficacy of intravenous remimazolam in inducing and maintaining suitable sedation levels for paediatric patients undergoing diagnostic and/or therapeutic procedures

DETAILED DESCRIPTION:
This trial is part of the European Paediatric Investigational Plan and the US Pediatric Study Plan and has been developed in line with guidance from the EMA Paediatric Committee and the US FDA.

The trial will commence with cohort 1 (aged ≥6 and <18 years) and proceed to lower age groups: cohort 2 (≥3 and <6 years); and, in European sites only, cohort 3 (full-term birth to <3 years). The Data Monitoring committee (DMC) may convene any time after at least half of the subjects in cohort 1 or 2 have completed the study, to review PK,safety and efficacy data. If there are no concerns, the DMC may recommend to initiate concurrent dosing in the next younger cohort (cohort 2 or 3) in parallel to dosing the remaining subjects in cohort 1 or 2 Dosing for cohort 3 will be predicted based on PK modelling as well as efficacy and safety outcomes of the older age groups. Enrolment of patients aged <2 years will not be permitted until supported by adequate juvenile toxicity data.

The trial will consist of three visits: Screening (Day -21 to day 1),Treatment (Day 1), and Follow-up (Day 4 [+3/-1 days]).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form and/or assent and willingness of patient and parent(s) to participate in the trial.
* In US sites: Paediatric male or female patients, aged ≥3 and <18 years scheduled to undergo a diagnostic or therapeutic procedure, which is medically indicated and independent from the trial.
* In European sites: Paediatric male or female patients, aged full term birth to <18 years scheduled to undergo a diagnostic or therapeutic procedure, which is medically indicated and independent from the trial.
* Maximum planned duration of procedure: 2 hours
* ASA Physical Status I-III
* Planned spontaneous breathing during sedation
* A female who is of child bearing potential (i.e. after menarche) and sexually active must use a highly effective method of birth control during the trial period (from the time of consent until all specified observations are completed)
* Negative pregnancy test at screening and on treatment day -

Exclusion Criteria:

* Emergency procedures
* Condition/procedure that requires planned airway control via endotracheal tube or LMA/IGEL insertion
* Cranio-facial malformation, which would severely limit the possibilities for emergency airway rescue
* Other abnormalities relating to the airway (including large tonsils and anatomical abnormalities of upper airway or lower airway) which may compromise emergency airway rescue
* Known hypersensitivity to benzodiazepines, flumazenil, dextran or any of the ingredients of the drug product
* Known paradoxical reactions to benzodiazepines
* History of sleep apnoea
* Active respiratory failure
* Active neuromuscular disease
* Active cardiac failure
* Active hepatic failure
* Breast feeding females
* Prohibited medication
* Any patient judged by the Principal Investigator (PI) or Sub-Investigator to be inappropriate for the trial for any other reason

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Success of the procedure | 2 hours
  Success of the procedure defined as: Completion of the procedure AND no requirement for rescue sedative medication AND no requirement for more than the permitted bolus or infusion regimen

SECONDARY OUTCOMES:
Target depth of sedation achieved | 2 hours
  Proportion of patients achieving predefined target depth of sedation (assessed using University of Michigan Sedation Score [UMSS]) during procedure
Target range of sedation achieved during 80% of procedure duration | 2 hours
  Proportion of patients in whom predefined target range of sedation (assessed using University of Michigan Sedation Score [UMSS]) was achieved during at least 80% of procedure duration
Percentage of time within target range of sedation | 2 hours
  Percentage of time spent by patients within predefined target range of sedation (assessed using University of Michigan Sedation Score [UMSS]) during procedure
Adequacy of sedation | 2 hours
  Depth of sedation (assessed using Nurse Interpretation of Sedation Scale [NISS]) of patients over time
Time to start of procedure | 2 hours
  Time between initial administration of study drug and start of procedure
Time to fully alert | 2 hours
  Time between last dose of study drug, end of procedure and full alertness, defined as the first of three consecutive sedation scores showing no sedation
Time to ready for discharge | 2 hours
  Time between last dose of study drug, end of procedure and discharge readiness
Signs of re-sedation | 2 hours
  Occurrence, after reaching a University of Michigan Sedation Score (UMSS) of 0 after end of procedure, of a UMSS greater than zero
Procedure success excluding cases where the procedure could not be completed for non sedative reasons | 2 hours
  Success of the procedure defined as: Completion of the procedure AND no requirement for rescue sedative medication AND no requirement for more than the permitted bolus or infusion regimen; excluding any patients where procedure was not completed for reasons other than failure of sedation
Safety: AEs | 4 days
  Incidence of treatment-emergent adverse events
Safety: emergence of delirium | 2 hours
  Incidence of paediatric anaesthesia emergence delirium between end of procedure until fit for discharge
Safety: need for ventilation | 2 hours
  Incidence of use of any manual or mechanical ventilation
Safety: need for reversal | 2 hours
  Incidence of use of flumazenil for reversal of benzodiazepine effect
PK: assessment of plasma concentration-time relationship | 3.5 hours
  Graphical description of plasma concentration over time and comparison to predicted concentration-time relationship as calculated from existing pharmacokinetic/pharmacodynamic model

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - Stanford University, Palo Alto, California
  - University of California Davis Children's Hospital, Sacramento, California
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - University of Pittsburgh Medical Center - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Odense Universitetshospital, Odense

IPD SHARING:
Plan to Share IPD: No